CLINICAL TRIAL: NCT02157116
Title: Dose-Dense Induction/Neoadjuvant Chemotherapy in the Treatment of Patients With Locally Advanced Non-Small Cell Lung Cancer With Additional Genomic Analyses to Identify Signatures Predictive of Chemotherapy Response.
Brief Title: Dose-Dense Induction/Neoadjuvant Chemotherapy in Locally Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual to meet analysis goals
Sponsor: Duke University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004682
Record Dates: First submitted 2014-05-29; First posted 2014-06-05 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Dose-Dense Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction Chemotherapy (Experimental): Cisplatin 75mg/m2 IV days 1, 15, 29; Docetaxel 75mg/m2 IV days 1, 15, 29; and Pegfilgrastim 6mg SC day 2, 16, 30
  Interventions: Drug: cisplatin; Drug: Docetaxel; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: cisplatin
  Other Names: Platinol
Drug: Docetaxel
  Other Names: Taxotere
Drug: Pegfilgrastim
  Other Names: Neulasta

SUMMARY:
Dose-dense chemotherapy is a chemotherapy treatment plan in which drugs are given with less time between treatments than in standard chemotherapy. The two chemotherapy drugs used in this study, docetaxel and cisplatin, are approved for the treatment of lung cancer when given every 21 days. This study is exploring the response to chemotherapy when these drugs are given every 14 days. In addition, genetic tests will be performed on pre-treatment specimens to identify signatures that may predict chemotherapy sensitivity or resistance.

DETAILED DESCRIPTION:
All patients will receive induction chemotherapy with cisplatin and docetaxel. Pegfilgrastim will be administered approximately 24 hours following the end of the day 1 chemotherapy infusion. Cycles will be repeated every 2 weeks for 3 cycles. Patients deemed to be resectable will undergo surgical resection followed by postoperative thoracic radiotherapy. Patients deemed inoperable will additionally receive concurrent chemoradiotherapy. Response, using radiographic and/or pathologic means, will identify two cohorts; responders and nonresponders.Gene expression profiling will then be performed on pre-treatment specimens to identify signatures that predict for chemotherapy sensitivity or resistance.

The target enrollment is 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented stage III NSCLC (IIIA or IIIB, without malignant pleural/pericardial effusion) are eligible for enrollment if they are considered appropriate for treatment with chemotherapy, radiation, or surgery;
* IIIA: T1-3 N2 M0, T3 N1 M0
* IIIB: T4 N0-2 M0, T 1-4 N3 M0
* Measurable or evaluable disease
* Previously untreated with chemotherapy or radiotherapy for lung cancer;
* No brain metastases;
* No prior XRT
* Performance status 0-2
* ≥18 years of age
* Informed Consent
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Bilirubin ≤ 1.5 x upper limit of normal for the institution (ULN)
* SGOT and SGPT ≤ 2.5 x ULN for the institution
* Creatinine ≤ 1.6 mg/dL
* Hemoglobin ≥ 8.0 g/dL
* Peripheral neuropathy ≤ grade 1

Exclusion Criteria:

* Known sensitivity to E. coli derived products (e.g. Filgrastim, HUMULIN® insulin, L-asparaginase, HUMATROPE® Growth Hormone, INTRON® A);
* Use of IV systemic antibiotics within 72 hours prior to chemotherapy;
* Known HIV infection
* Lithium or cytokines within 2 weeks prior of entry
* Additional concurrent investigational drugs
* History of myelodysplastic syndrome
* Pregnant, nursing or having unprotected sex
* Not available for follow-up assessment
* Unable to comply with protocol procedures
* Illnesses that may compromise ability to give informed consent.
* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to enrollment in May 2006 and closed in October 2009 due to failure to meet accrual goals for data analysis.
Groups:
- All Subjects: All subjects who signed a consent form are included, whether or not they received treatment as a part of the study.
Period: Overall Study
Arm/Group | All Subjects
Started | 13 (signed consent form)
Completed | 4
Not Completed | 9
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 3
Not completed — Failed Screening | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 13
Age, Customized [Number; unit: years]
  <18 years | 0
  >= 18 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Induction Response
Description: Response will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Response is defined as the number patients with a Complete Response (CR), disappearance of all target lesions, or a Partial Response (PR), at least a 30% decrease in the sum of the longest diameter (LD) of target lesions.
Time Frame: Between 2 and 3 weeks after induction
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Differential Gene Expression Between Responsive and Resistant Tumor Treated With Dose-dense Therapy
Time Frame: at the end of the study, estimated 2.5 years
Population: Due to insufficient accrual, gene analysis was not performed.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Grade III/IV Hematologic Adverse Events
Time Frame: During induction chemotherapy, approximately 6 weeks
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Grade III/IV Non-hematologic Adverse Events
Time Frame: During induction chemotherapy, approximately 6 weeks
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients Who Were Able to Maintain Hemoglobin Between 11-13 g/dL During Induction
Time Frame: During induction, approximately 6 weeks
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Time Frame: Approximately 10 years
Population: Due to insufficient accrual, the study was stopped prior to completing the 10 year followup for survival.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Treated Patients: Due to insufficient accrual, adverse event data was not analyzed.
Arm/Group | Treated Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No